CLINICAL TRIAL: NCT03492684
Title: Study of Superior Gluteal Mononeuropathy After Total Hip Arthroplasty Through Modified Direct Lateral Approach
Brief Title: Superior Gluteal Neuropathy -Total Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hamed Mohamed, DR.mohamed hamed, Assiut University
Other Study IDs: neuropathy - hip arthroplasty
Record Dates: First submitted 2018-03-23; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: ElectroPhys: Mononeuropathy
Keywords: nerve injury after total hip arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: total hip arthroplasty — total hip arthroplasty and EMG
  Other Names: electrophysiological study

SUMMARY:
A prospective study of 50 consecutive patients undergoing total hip arthroplasty, to establish whether there greater incidence of injury to the superior gluteal nerve associated with a particular approach (modified direct lateral approach). The patients will be assessed clinically and electrophysiologically before and after the operation through one year.

DETAILED DESCRIPTION:
Neurological complications following total hip arthroplasty are uncommon, and their impact ranges from transient and trivial to permanent and devastating.

In general, the prevalence rate of neurologic injury after primary hip arthroplasty is estimated as 0.7-3.5% , whereas it may increase up to 7.6% after revision hip arthroplasty.

Direct or indirect injuries of nerves may occur during operative exposure and subsequent procedures. Injuries to the peripheral nerves can come about in several ways: laceration, ischemia, mechanical deformation from compression or distraction, or a combination of these causes.

Peripheral nerve injuries can involve either distant sites or nerves in the immediate vicinity of the hip joint. Sciatic nerve injury is the most common nerve to be injured following total hip arthroplasty. Femoral nerve injury is much less common and is associated with an anterior approach. Its diagnosis is often delayed, but the prognosis is generally better than with sciatic nerve injury.

The direct lateral approach to the hip was described by Hardinge and is based on the observation that the gluteus medius and vastus lateralis are in functional continuity through the thick tendinous periosteum covering the greater trochanter.

This approach involves splitting the gluteus medius and retracting a portion of the muscle anteriorly in continuity with part of the vastus lateralis. It avoids trochanteric osteotomy, but the neurovascular supply of gluteus medius and tensor fascia lata is vulnerable.

The superior gluteal nerve may be compromised during total hip arthroplasty done through the direct lateral approach of Hardinge which puts this nerve at risk when the gluteus medius is split and retracted anteriorly.

The function of the abductors may be impaired after operation if there is damage to the superior gluteal nerve or if the muscle flap is reattached inadequately to the trochanter.

ELIGIBILITY:
Inclusion Criteria:

* Age: adults
* Sex: both males and female
* Operation: unilateral primary total hip replacement

Exclusion Criteria:

* Patient refusal
* Patients with pre-existing neuromuscular abnormality
* Preoperative immobility
* patient with bilateral total hip arthroplasty or hip pathology
* Revision hip arthroplasty

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Age: adults
  * Sex: both males and female
  * Operation: unilateral primary total hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with failure of initial intervention | one year
  prospective case series study study of Superior gluteal mononeuropathy after total hip arthroplasty through modified direct lateral approach by EMG studies

CONTACTS AND LOCATIONS:
Overall Officials: mohamed hamed mohamed, Principal Investigator — Assiut University

REFERENCES:
- [Background] Edwards BN, Tullos HS, Noble PC. Contributory factors and etiology of sciatic nerve palsy in total hip arthroplasty. Clin Orthop Relat Res. 1987 May;(218):136-41. PMID 3568473
- [Background] Yang IH. Neurovascular Injury in Hip Arthroplasty. Hip Pelvis. 2014 Jun;26(2):74-8. doi: 10.5371/hp.2014.26.2.74. Epub 2014 Jun 30. PMID 27536562
- [Background] Solheim LF, Hagen R. Femoral and sciatic neuropathies after total hip arthroplasty. Acta Orthop Scand. 1980 Jun;51(3):531-4. doi: 10.3109/17453678008990836. PMID 6255726
- [Background] Schmalzried TP, Amstutz HC, Dorey FJ. Nerve palsy associated with total hip replacement. Risk factors and prognosis. J Bone Joint Surg Am. 1991 Aug;73(7):1074-80. PMID 1874771